CLINICAL TRIAL: NCT05232851
Title: Stimulating Immune Response With Neoadjuvant Human Papilloma Virus (HPV)-16 Specific Vaccination in HPV-Oropharyngeal Squamous Cell Carcinoma (HPV-OPSCC)
Brief Title: A Vaccine (PDS0101) Alone or in Combination With Pembrolizumab for the Treatment of Locally Advanced Human Papillomavirus-Associated Oropharynx Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MC200710; NCI-2022-00497 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-006302 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Human Papillomavirus-Related Carcinoma; Locally Advanced Oropharyngeal Carcinoma; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Carcinoma | interventions — pembrolizumab; Specimen Handling; Biopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Pathologist will be blinded to study treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (PDS0101) (Experimental): Patients receive PDS0101 SC on day 1 of each cycle. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or FDG-PET/CT and blood sample collection throughout the trial. Patients may undergo a biopsy during screening and on the trial.
  Interventions: Biological: Liposomal HPV-16 E6/E7 Multipeptide Vaccine PDS0101; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography; Procedure: Biospecimen Collection; Procedure: Biopsy
- Arm B (PDS0101, pembrolizumab) (Experimental): Patients receive PDS0101 SC on day 1 and pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or FDG-PET/CT and blood sample collection throughout the trial. Patients may undergo a biopsy during screening and on the trial.
  Interventions: Biological: Liposomal HPV-16 E6/E7 Multipeptide Vaccine PDS0101; Biological: Pembrolizumab; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography; Procedure: Biospecimen Collection; Procedure: Biopsy

INTERVENTIONS:
Biological: Liposomal HPV-16 E6/E7 Multipeptide Vaccine PDS0101 — Given SC
  Other Names: mmunoMAPK-RDOTAP /HPV-16 E6/E7 Peptide Antigen Vaccine; PDS0101
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Biosimilar BCD-201; Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Arm B (PDS0101, pembrolizumab)
Procedure: Computed Tomography — Undergo CT, FDG-PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography; CT; CT SCAN; tomography
Procedure: FDG-Positron Emission Tomography — Undergo FDG-PET/CT
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx

SUMMARY:
This phase I/II trial studies how well PDS0101 alone or in combination with pembrolizumab works to shrink tumor in patients with human papillomavirus-associated oropharynx cancer that has spread to nearby tissue or lymph nodes (locally advanced). PDS0101 is a vaccine made from specific peptides that may help the body build an effective immune response to kill tumor cells. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving PDS0101 with or without pembrolizumab may kill more tumor cells in patients with locally advanced human papillomavirus-associated oropharynx cancer before surgery so that it may make the tumor smaller and may reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine pathologic and human papillomavirus cell-free tumor deoxyribonucleic acid (ctHPVDNA) response to liposomal HPV-16 E6/E7 multipeptide vaccine PDS0101 (PDS0101) or PDS0101 plus pembrolizumab in patients with high risk human papillomavirus-associated oropharynx cancer (HPV-OPSCC).

SECONDARY OBJECTIVES:

I. To determine tumor response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

II. To determine progression-free survival and overall survival.

TERTIARY OBJECTIVES:

I. To determine the safety of PDS0101 delivered alone or with pembrolizumab.

CORRELATIVE RESEARCH OBJECTIVES:

I. Determine the changes in tumor microenvironment (TME) with PDS0101 alone or with pembrolizumab.

II. Determine circulating ctHPVDNA as a biomarker for tumor response. III. Determine HPV16-specific T-cell response utilizing multiplex flow cytometry and other parameters.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive PDS0101 subcutaneously (SC) on day 1 of each cycle. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/CT and blood sample collection throughout the trial. Patients may undergo a biopsy during screening and on the trial.

ARM B: Patients receive PDS0101 SC on day 1 and pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or FDG-PET/CT and blood sample collection throughout the trial. Patients may undergo a biopsy during screening and on the trial.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Disease characteristics

  * Locally advanced HPV-OPSCC and high-risk HPV-specific testing with at least one of the following:

    * Radiology extranodal extension (ENE) OR
    * cN2 (AJCC 8th Edition) disease (contralateral/bilateral nodes) OR
    * cN3(AJCC 8th Edition) disease (lymph node [LN] > 6 cm) OR
    * Radiographic evidence of 2 or more involved lymph nodes
  * Candidate for curative intent surgery or chemo-radiation
* Measurable or unmeasurable disease as defined by RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* White blood cell (WBC) count >= 3,000/mm^3 (=< 15 days prior to registration)
* Platelet count >= 75,000/mm^3 (=< 15 days prior to registration)
* Hemoglobin >= 9.0 g/dL (5.6 mmol/L) (=< 15 days prior to registration)

  * NOTE: Transfusions are not allowed =< 7 days prior to registration
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (or total bilirubin =< 3.0 X ULN with direct bilirubin =<1.5 X ULN in patients with well-documented Gilbert's Syndrome) (=< 15 days prior to registration)
* Aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/SGOT) =< 2.5 X ULN (=< 15 days prior to registration)
* Creatinine =< 1.5 mg/dL (133 umol/L) OR calculated creatinine clearance >= 30 mL/min/1.73m^2 for patients with creatinine levels above ULN (=< 15 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.5 X ULN OR if patient is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of anticoagulants (=< 15 days prior to registration)
* Negative pregnancy test done =< 3 days prior to registration for persons of childbearing potential only
* Persons of childbearing potential or able to father a child must be willing to use an effective method of contraception for the course of the study starting with the first dose of study therapy through 120 days after the last dose of study medication

  * NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred method of contraception for the patient
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research

Exclusion Criteria:

* Active autoimmune disease requiring systemic treatment, documented history of severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents

  * NOTE: Exceptions are allowed for:

    * Vitiligo
    * Resolved childhood asthma/atopy
    * Intermittent use of bronchodilators or inhaled steroids
    * Daily steroids at dose of =< 10mg of prednisone (or equivalent)
    * Local steroid injections
    * Stable hypothyroidism on replacement therapy
    * Stable diabetes mellitus
    * Sjogren's syndrome
* Any prior head or neck chemotherapy, radiotherapy, and/or immunotherapy
* Any of the following prior therapies:

  * Live vaccine < 30 days prior to registration, including intranasal flu vaccine (e.g. Flu-Mist®) (Note: Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed). Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist) are live attenuated vaccines and are not allowed
  * Chemotherapy or targeted small molecule therapy < 21 days prior to registration
  * Investigational therapy or investigational device < 30 days prior to registration
  * Any prior investigational HPV-specific therapeutic vaccine
* Current or prior use of immunosuppressive medication < 14 days prior to registration

  * The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intraarticular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., premedication for computed tomography [CT] scans)
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic therapy
  * Interstitial lung disease
  * Serious, chronic gastrointestinal conditions associated with diarrhea (e.g., Crohn's disease or others)
  * Known active hepatitis B (i.e., known positive HBV surface antigen (HBsAg) reactive)
  * Known active hepatitis C (i.e., positive for HCV ribonucleic acid [RNA] detected by polymerase chain reaction [PCR])
  * Known human immunodeficiency virus (HIV) (Note: Patients on stable highly active antiretroviral therapy (HAART) for >= 6 weeks with CD4 counts >= 200 cells/mm^3 undetectable HIV viral load by quantitative PCR and no opportunistic infections Castlemaan's Disease =< 12 months prior to enrollment are allowed)
  * Known active tuberculosis (TB)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Unstable cardiac arrhythmia or
  * Psychiatric illness/social situations that would limit compliance with study requirements (e.g., substance abuse)
* History of allogeneic hematopoietic transplant or any solid organ transplant
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy < 2 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer (SCC/BCC), micropapillary thyroid cancer, Gleason 6 prostate cancer, carcinoma-in-situ of the breast or cervix
* Any of the following conditions =< 6 weeks prior to registration:

  * Cerebrovascular accident (CVA)
  * Admission for unstable angina
  * Cardiac angioplasty or stenting or coronary artery bypass graft surgery
  * Untreated pulmonary embolism or untreated deep venous thrombosis (DVT)
  * Arterial thrombosis
* Receipt of immunotherapy/immunomodulatory or immunosuppressive agents (e.g., IFNs, tumor necrosis factor, interleukins, immunoglobulins or other biologic response modifiers [GM-CSF, GCSF] =< 6 weeks prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Proportion of pathologic and human papillomavirus cell-free tumor deoxyribonucleic acid (ctHPVDNA) response | Up to 2 years
  Will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the exact binomial method for each arm separately.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From registration to the first of either disease progression or death from any cause, assessed up to 2 years
  Patients who receive the study drug, but then never return for an evaluation will be censored on their last follow-up date. PFS will be estimated using the method of Kaplan-Meier. PFS rates at 12 and 24 months will also be reported.
Overall survival (OS) | From registration to death from any cause, assessed up to 2 years
  OS will be estimated using the method of Kaplan Meier.
Response rate | Up to 2 years
  Will be estimated using Response Evaluation Criteria in Solid Tumors 1.1 criteria. A tumor response is defined to be either a complete response or partial response noted up until surgery. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response. Patients who go off study early before having a tumor assessment performed will be considered a failure.
Incidence of adverse events (AEs) | Up to 30 days after treatment discontinuation
  All patients that have initiated treatment will be considered evaluable for AE analyses. The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine AE patterns. AEs will be analyzed separately by arm.

CONTACTS AND LOCATIONS:
Overall Officials: David M. Routman, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials